CLINICAL TRIAL: NCT03773302
Title: A Phase 3 Multicenter, Open-Label, Randomized, Controlled Study of Oral Infigratinib Versus Gemcitabine With Cisplatin in Subjects With Advanced/Metastatic or Inoperable Cholangiocarcinoma With FGFR2 Gene Fusions/Translocations: The PROOF Trial
Brief Title: Phase 3 Study of BGJ398 (Oral Infigratinib) in First Line Cholangiocarcinoma With FGFR2 Gene Fusions/Translocations
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The sponsor has decided to close the study due to the discontinuation of infigratinib development in oncology within the sponsor's territory. The discontinuation of the study was not due to safety issues.
Sponsor: QED Therapeutics, a BridgeBio company (Industry)
Collaborators: Helsinn Healthcare SA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: QBGJ398-301; 2018-004004-19 (EudraCT Number)
Record Dates: First submitted 2018-12-10; First posted 2018-12-12 (Actual); Results first posted 2024-05-08 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-04

CONDITIONS: Advanced Cholangiocarcinoma; FGFR2 Gene Mutation
Keywords: cholangiocarcinoma; unresectable cholangiocarcinoma; metastatic cholangiocarcinoma; fibroblast growth factor receptor inhibitor; FGFR2; FGFR2 gene fusions/translocations; BGJ398
MeSH Terms: conditions — Cholangiocarcinoma | interventions — infigratinib; Gemcitabine; Cisplatin

STUDY DESIGN:
Intervention Model Description: Multicenter, Open Label, 2:1 Randomized, Controlled Phase 3
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Infigratinib (BGJ398) 125 mg (Experimental): Infigratinib (BGJ398) 125 mg orally daily, 3 weeks on, 1 week off.
  Interventions: Drug: BGJ398
- Gemcitabine + Cisplatin (Active Comparator): Participants who experience disease progression while receiving gemcitabine + cisplatin will be allowed to cross over and receive infigratinib if certain criteria are met.
  Interventions: Drug: Gemcitabine; Drug: Cisplatin

INTERVENTIONS:
Drug: BGJ398 — Infigratinib (BGJ398) 125 mg orally daily, 3 weeks on, 1 week off.
  Other Names: Infigratinib
  Arms: Infigratinib (BGJ398) 125 mg
Drug: Gemcitabine — Gemcitabine 1000 mg/m2 IV D1 and D8 for a 21-day cycle. Participants who experience disease progression while receiving gemcitabine + cisplatin will be allowed to cross over and receive infigratinib.
  Arms: Gemcitabine + Cisplatin
Drug: Cisplatin — Cisplatin 25 mg/m2 IV D1 and D8 for a 21-day cycle. Participants who experience disease progression while receiving gemcitabine + cisplatin will be allowed to cross over and receive infigratinib.
  Arms: Gemcitabine + Cisplatin

SUMMARY:
Infigratinib is an oral drug which selectively binds to fibroblast growth factor receptor (FGFR) 2 and is being developed to treat participants with FGFR2 mutated cholangiocarcinoma. The purpose of the study is to evaluate the efficacy and safety of the investigational agent oral infigratinib vs standard of care chemotherapy (gemcitabine plus cisplatin) in first-line treatment of participants with unresectable locally advanced or metastatic cholangiocarcinoma with FGFR2 fusion/rearrangement. Subjects will be randomized 2:1 to receive infigratinib or gemcitabine plus cisplatin.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed unresectable locally advanced or metastatic cholangiocarcinoma. Participants with gallbladder cancer or ampulla of Vater carcinoma are not eligible
* Have written documentation of local laboratory or central laboratory determination of a known or likely activating FGFR2 fusion/rearrangement from a sample collected before randomization
* Have an archival tumor tissue sample available with sufficient tumor content for FGFR2 fusion/rearrangement molecular testing by the central laboratory. However, if an archival tumor tissue sample is not available, or does not meet requirements for central testing a newly obtained (before randomization) tumor biopsy may be submitted instead. If a prestudy written documentation of FGFR2 fusion/rearrangement in tumor tissue is available from the central laboratory, an additional tumor sample does not need to be submitted.
* Have an Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1
* Are able to swallow and retain oral medication
* Are willingness to avoid pregnancy or father children

Exclusion Criteria:

* Received treatment with any systemic anti-cancer therapy for unresectable locally advanced or metastatic cholangiocarcinoma, with following exceptions

  1. Prior neoadjuvant or adjuvant therapy is permitted if completed > 6 months after the last dose of neoadjuvant or adjuvant therapy.
  2. One cycle of gemcitabine-based chemotherapy for locally advanced or metastatic cholangiocarcinoma is permitted before randomization
* History of a liver transplant
* Received previously or currently is receiving treatment with a mitogen activated protein kinase kinase (MEK) or selective FGFR inhibitor
* Have impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of oral infigratinib (such as, ulcerative diseases, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome, small bowel resection).
* Current evidence of endocrine alterations of calcium/phosphate homeostasis, e.g., parathyroid disorders, history of parathyroidectomy, tumor lysis, tumoral calcinosis etc.
* History and/or current evidence of extensive tissue calcification including, but not limited to, the soft tissue, kidneys, intestine, myocardium, vascular system and lung with the exception of calcified lymph nodes, minor pulmonary parenchymal calcifications, and asymptomatic coronary calcification
* Current evidence of corneal or retinal disorder/keratopathy
* Receiving and continued treatment or are planning to receive agents or consuming foods that are known moderate or strong inducers or inhibitors of CYP3A4 and medications which increase serum phosphorus and/or calcium concentration
* Clinically significant or uncontrolled cardiac disease
* Recent (≤ 3 months prior to first dose of study drug) transient ischemic attack or stroke
* Severe hearing loss
* Severe neuropathy
* History of another primary malignancy within 3 years except adequately treated in-situ carcinoma of the cervix or non-melanoma skin cancer or other curatively treated malignancy that is not expected to require treatment
* Pregnant or breastfeeding
* Have known microsatellite instability-high (MSI-H) disease and the decision is made by the treating investigator that an alternative, non-study therapy is warranted according to standard of care.
* Have any known hypersensitivity to gemcitabine, cisplatin, calcium-lowering agents, infigratinib, or their excipients
* Have any contraindication to cisplatin or gemcitabine treatment according to local labeling or standard institutional practice.
* Have taken any Chinese herbal medicine or Chinese patent medicine treatments with anticancer activity within 14 days of the first dose of study drug.
* Have received a live vaccine within 30 days before the first dose of study drug or are planning to receive a live vaccine during participation in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2019-12-27 (Actual); Primary Completion 2023-03-02 (Actual); Study Completion 2023-03-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Development, Study Director — QED Therapeutics
Locations (116):
- United States (25):
  - Banner MD Anderson Cancer Center, Gilbert, Arizona
  - University of Arizona, Tucson, Arizona
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - St. Joseph Heritage Healthcare, Fullerton, California
  - USC Norris Cancer Center, Los Angeles, California
  - University of California Los Angeles, Los Angeles, California
  - Florida Hospital Medical Group, Orlando, Florida
  - UF Health Cancer Center at Orlando Health, Orlando, Florida
  - Northwestern Memorial Hospital, Chicago, Illinois
  - University Medical Center - New Orleans, New Orleans, Louisiana
  - Frederick Regional Healthcare Systems/James M. Stockman Cancer Institute, Frederick, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Barbara Ann Karmanos Cancer Institute - Lawrence and Idell Weisberg Cancer Treatment Center, Detroit, Michigan
  - Cancer and Hematology Centers of Western Michigan, Grand Rapids, Michigan
  - William Beaumont Hospital, Royal Oak, Michigan
  - NYU Langone Medical Center, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Levine Cancer Institute - Charlotte, Charlotte, North Carolina
  - University of Cincinnati Medical Center, Cincinnati, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Charleston Oncology, Charleston, South Carolina
  - Parkland Health and Hospital System, Dallas, Texas
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - University of Texas MD Anderson Cancer Center, Houston, Texas
  - Baylor College of Medicine, Houston, Texas
- Australia (6):
  - Chris O'Brien Lifehouse Hospital, Camperdown, New South Wales
  - Blacktown Hospital, Darlinghurst, New South Wales
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Monash Medical Centre, Bentleigh East, Victoria
  - Peninsula & South Eastern Haematology and Oncology Group, Frankston, Victoria
  - St John of God Hospital Subiaco, Subiaco, Western Australia
- Belgium (3):
  - Cliniques Universitaires Saint-Luc, Brussels, Brussels Capital
  - Grand Hopital de Charleroi, Charleroi
  - Universitair Ziekenhuis Antwerpen, Edegem
- Canada (4):
  - Cross Cancer Institute, Edmonton, Alberta
  - Ottawa Hospital, Ottawa, Ontario
  - St. Josephs Health Centre, Toronto, Ontario
  - Jewish General Hospital, Montreal, Quebec
- China (8):
  - Peking University People's Hospital, Beijing
  - Beijing Cancer Hospital, Beijing
  - Peking University Third Hospital, Beijing
  - Hunan Cancer Hospital, Changsha
  - Guangzhou First People's Hospital, Guangzhou
  - Hubei Cancer Hospital, Hubei
  - Liaoning Cancer Hospital & Institute, Shenyang
  - The First Affiliated Hospital, Sun Yat-sen University, Zhongshan
- France (10):
  - Hopital Henri Mondor, Créteil, Val-de-Marne
  - CHRU Dijon, Dijon
  - Centre Georges-Francois Leclerc, Dijon
  - Hopital Claude Huriez Rue Michel Polonovski (CHRU) Lille, Lille
  - Groupement Hospitalier Edouard Herriot, Lyon
  - Hopital Nord Franche-Comte, Montbéliard
  - Groupe Hospitalier Archet I Et II, Nice
  - Hopital Cochin, Paris
  - Hôpital Saint Antoine, Paris
  - L'Institut Mutualiste Montsouris, Paris
- Germany (4):
  - Universitätsklinikum Tübingen, Tübingen, Baden-Wurttemberg
  - Klinikum rechts der Isar der Technischen Universität München, München, Bavaria
  - Klinikum Dortmund gGmbH, Dortmund
  - University Clinic Heidelberg, Heidelberg
- Italy (6):
  - Azienda Socio Sanitaria Territoriale di Cremona (ASST), Cremona
  - Istituto Scientifico Romagnolo Per Lo Studio E La Cura Dei Tumori IRST, Meldola
  - Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico, Milan
  - ASST Grande Ospedale Metropolitano Niguarda, Milan
  - Istituto Oncologico Veneto - I.R.C.C.S., Padua
  - Policlinico Universitario Campus Biomedico Di Roma, Roma
- Portugal (10):
  - Hospital Beatriz Angelo, Loures, Lisbon District
  - Hospital Garcia de Orta, Almada
  - Centro Hospitalar E Universitário de Coimbra EPE, Coimbra
  - Instituto Português de Oncologia Francisco Gentil Centro Regional de Oncologia de Coimbra EPE, Coimbra
  - Instituto Português de Oncologia de Lisboa Francisco Gentil, E.P.E., Lisbon
  - Centro Hospitalar Lisboa Norte, E.P.E. - Hospital de Santa Maria, Lisbon
  - Hospital CUF Descobertas, Lisbon
  - Centro Hospitalar do Porto - Hospital de Santo António, Porto
  - Instituto Portugues de Oncologia Do Porto Francisco Gentil Epe - PPDS, Porto
  - Centro Hospitalar de São João, E.P.E., Porto
- Hospital Oncologico, Puerto Rico Medical Center, Rio Piedras, Puerto Rico
- South Korea (8):
  - Pusan National University Hospital, Pusan
  - Seoul National University Bundang Hospital, Seongnam-si
  - SMG - SNU Boramae Medical Center, Seoul
  - Samsung Medical Center, Seoul
  - Seoul National University Hospital, Seoul
  - Severance Hospital Yonsei University Health System, Seoul
  - The Catholic University of Korea, Seoul St. Mary's Hospital, Seoul
  - Ajou University Hospital, Suwon
- Spain (12):
  - Hospital Universitario Virgen Macarena, Seville, Andalusia
  - Hospital Universitario Miguel Servet, Zaragoza, Aragon
  - Complejo Asistencial Universitario de Salamanca - Hospital Clinico, Salamanca, Castille and León
  - Hospital Universitario Germans Trias i Pujol, Badalona, Catalonia
  - Instituto Catalan de Oncologio ICO I'Hospitalet, Barcelona, Catalonia
  - Hospital Universitario Vall d'Hebrón - PPDS, Barcelona
  - Hospital General Universitario Gregorio Maranon, Madrid
  - Hospital Universitario Ramon y Cajal, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario HM Sanchinarro - CIOCC, Madrid
  - Hospital Universitari i Politecnic La Fe de Valencia, Valencia
- Taiwan (8):
  - National Cheng Kung University Hospital, Tainan, Tainan
  - National Taiwan University Hospital - YunLin Branch, Huwei
  - Chang Gung Memorial Hospital - Kaohsiung, Kaohsiung City
  - China Medical University Hospital, Taichung
  - Chi Mei Hospital, Liouying, Tainan
  - Taipei Veterans General Hospital, Taipei
  - National Taiwan University Hospital, Taipei
  - Chang Gung Memorial Hospital, Linkou, Taoyuan
- Thailand (6):
  - Songklanagarind Hospital, Prince of Songkla University, Hat Yai, Changwat Songkhla
  - Chulalongkorn University, Bangkok
  - Ramathibodi Hospital Mahidol University, Bangkok
  - Maharaj Nakorn Chiang Mai Chiang Mai University, Chiang Mai
  - Srinagarind Hospital, Khon Kaen
  - Naresuan University, Phitsanulok
- United Kingdom (5):
  - Nottingham City Hospital, Nottingham, Nottinghamshire
  - Royal Marsden Hospital, Sutton, Surrey
  - The Clatterbridge Cancer Centre NHS Foundation Trust, Bebington, Wirral
  - Guys Hospital, London
  - The Christie NHS Foundation Trust - PPDS, Manchester

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Makawita S, K Abou-Alfa G, Roychowdhury S, Sadeghi S, Borbath I, Goyal L, Cohn A, Lamarca A, Oh DY, Macarulla T, T Shroff R, Howland M, Li A, Cho T, Pande A, Javle M. Infigratinib in patients with advanced cholangiocarcinoma with FGFR2 gene fusions/translocations: the PROOF 301 trial. Future Oncol. 2020 Oct;16(30):2375-2384. doi: 10.2217/fon-2020-0299. Epub 2020 Jun 25. PMID 32580579

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants with a diagnosis of advanced/metastatic or inoperable cholangiocarcinoma (CCA) with FGFR2 fusion/rearrangement were recruited to this open-label, randomized, controlled global study across Western Europe, North America, and Asia, based on documented evidence of FGFR2 genetic alteration. The first participant was treated on 18 March 2020. The data cutoff for the analysis was 02 March 2023.
Pre-assignment Details: Subjects meeting inclusion/exclusion criteria were randomly assigned 2:1 to receive oral infigratinib 125 mg (N=29) or gemcitabine+cisplatin (N=19). Randomization was stratified by unresectable locally advanced vs metastatic disease, geographic region (North America, Western Europe, Asia Pacific, and rest of the world), prior neoadjuvant/adjuvant treatment (yes/no) and received up to 1 cycle of prior gemcitabine-based chemotherapy for unresectable locally advanced or metastatic disease (yes/no).
Groups:
- Gemcitabine + Cisplatin: Gemcitabine: Gemcitabine 1000 mg/m2 IV D1 and D8 for a 21-day cycle.
  Cisplatin: Cisplatin 25 mg/m2 IV D1 and D8 for a 21-day cycle.
  Participants who experienced disease progression while receiving gemcitabine + cisplatin were allowed to cross over and receive infigratinib.
Period: Overall Study
Arm/Group | Infigratinib (BGJ398) 125 mg | Gemcitabine + Cisplatin
Started | 29 | 19 (Note: 2 subjects were randomized to the Gemcitabine/Cisplatin group but never received treatment.)
Completed | 29 | 17
Not Completed | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Gemcitabine + Cisplatin: Gemcitabine: Gemcitabine 1000 mg/m2 IV D1 and D8 for a 21-day cycle.
  Cisplatin: Cisplatin 25 mg/m2 IV D1 and D8 for a 21-day cycle.
- Total: Total of all reporting groups
Arm/Group | Infigratinib (BGJ398) 125 mg | Gemcitabine + Cisplatin | Total
Number analyzed (Participants) | 29 | 19 | 48
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 21 | 13 | 34
  >=65 years | 8 | 6 | 14
Age, Continuous [Mean (Standard Deviation); unit: years] | 54 (13.22) | 58.2 (15.25) | 55.8 (14.04)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 10 | 29
  Male | 10 | 9 | 19
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 7 | 3 | 10
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 20 | 14 | 34
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 2 | 3
Region of Enrollment [Number; unit: participants] — North America includes United States; Europe includes Belgium, Germany, and Spain; Asia includes Singapore, Thailand, and Taiwan.
  participants
    North America | 12 | 7 | 19
    Europe | 14 | 8 | 22
    Southeast Asia | 3 | 4 | 7
BMI [Mean (Standard Deviation); unit: kg/m2] | 28.41 (7.018) | 26.83 (8.019) | 27.79 (7.388)
ECOG PS [Count of Participants; unit: Participants] — Functional status was assessed at baseline using the Eastern Cooperative Oncology Group
  Performance Scale (ECOG PS), defined as follows:
  0. Fully active, able to carry out all pre-disease performance without restriction.
  1. Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature.
  2. Ambulatory and capable of all selfcare but unable to carry out any work activities; up and about more than 50% of waking hours.
  3. Capable of only limited selfcare; confined to bed or chair more than 50% of waking hours.
  4. Completely disabled.
  Participants
    0 | 19 | 8 | 27
    1 | 10 | 11 | 21
    2 | 0 | 0 | 0
Primary site of cholangiocarcinoma [Count of Participants; unit: Participants]
  Common bile duct | 1 | 1 | 2
  Intrahepatic bile duct | 28 | 17 | 45
  Other | 0 | 1 | 1
Histological subtype [Count of Participants; unit: Participants]
  Adenocarcinoma | 26 | 19 | 45
  Mixed adeno and squamous | 0 | 0 | 0
  Other | 3 | 0 | 3
Initial tumor (T) diagnosis category [Count of Participants; unit: Participants] — Tumor (T) TX: Main tumor cannot be measured. T0: Main tumor cannot be found. T1, T2, T3, T4: Refers to the size and/or extent of the main tumor. The higher the number after the T, the larger the tumor or the more it has grown into nearby tissues.
  Participants
    TX | 7 | 3 | 10
    T0 | 1 | 0 | 1
    Tis | 0 | 0 | 0
    T1 | 3 | 4 | 7
    T2 | 10 | 7 | 17
    T3 | 3 | 4 | 7
    T4 | 5 | 1 | 6
Initial metastasis (M) diagnosis category [Count of Participants; unit: Participants] — Distant metastasis (M) M0: Cancer has not spread to other parts of the body. M1: Cancer has spread to other parts of the body.
  Participants
    M0 | 8 | 5 | 13
    M1 | 21 | 14 | 35
    Missing | 0 | 0 | 0
Time from initial diagnosis to randomization [Mean (Standard Deviation); unit: months] | 8.49 (19.765) | 11.77 (20.582) | 9.79 (19.940)
FGFR2 Fusion - Local [Count of Participants; unit: Participants]
  Fusion positive - fusion partner known | 7 | 4 | 11
  Fusion positive - fusion partner unknown | 0 | 2 | 2
  Fusion positive - intron rearrangement | 2 | 2 | 4
  Fusion negative | 0 | 0 | 0
  Missing | 20 | 11 | 31
FGFR2 Fusion - Central [Count of Participants; unit: Participants]
  Fusion positive - fusion partner known | 15 | 10 | 25
  Fusion positive - fusion partner unknown | 2 | 0 | 2
  Fusion positive - intron rearrangement | 0 | 0 | 0
  Fusion negative | 0 | 0 | 0
  Missing | 12 | 9 | 21

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival (Central Imaging Assessment)
Description: Defined as the time from randomization until date of disease progression by blinded independent central imaging assessment (Response Evaluation Criteria in Solid Tumors [RECIST] v. 1.1) or death, whichever occurs first.
Time Frame: From the time of randomization to end of treatment due to confirmed disease progression or death. Note: PFS is an event driven endpoint. Subjects without confirmed disease progression at the end of study were censored at their last valid tumor assessment.
Measure: Median (Full Range); unit: Months
Arm/Group | Infigratinib (BGJ398) 125 mg | Gemcitabine + Cisplatin
Number analyzed (Participants) | 12 | 7
Months | 7.39 [0.03 to 12.85] | 8.02 [0.03 to 12.88]

2. Secondary Outcome: Overall Survival (OS) in Participants Treated With Infigratinib Versus Gemcitabine With Cisplatin
Description: OS by investigator assessment, defined as time from date of randomization until death due to any cause
Time Frame: From the time of randomization to time of death. Note: OS is an event driven endpoint. Subjects who had not died (no record of death) or were lost to follow-up were censored at the date of last known to be alive.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Infigratinib (BGJ398) 125 mg | Gemcitabine + Cisplatin
Number analyzed (Participants) | 8 | 3
Months | NA [14.36 to NA] — OS is an event driven endpoint. The number of events required to assess OS could not be calculated due to early termination of the study. | NA [8.02 to NA] — OS is an event driven endpoint. The number of events required to assess OS could not be calculated due to early termination of the study.

3. Secondary Outcome: Investigator Assessed Progression Free Survival in Participants Treated With Infigratinib Compared to Gemcitabine and Cisplatin
Description: Defined as the time from randomization until date of disease progression by site investigator (RECIST v1.1) or death, whichever occurs first.
Time Frame: as for outcome 1
Measure: Median (Full Range); unit: Months
Arm/Group | Infigratinib (BGJ398) 125 mg | Gemcitabine + Cisplatin
Number analyzed (Participants) | 19 | 8
Months | 7.39 [0.03 to 20.24] | 5.19 [0.03 to 12.88]

4. Secondary Outcome: Overall Response Rate (ORR) Determined by Blinded Independent Central (BICR) and Investigator Assessment
Description: ORR is defined as the proportion of subjects with a best overall response (BOR) of either confirmed partial response (PR) or confirmed complete response (CR) as assessed by BICR and the investigator according to RECIST v1.1 among patients with measurable disease at baseline
Time Frame: From the time of randomization to end of study treatment (an average of approx.6.5 months [max: 23 months] for the infigratinib arm and approx. 4 months [max: 11-13 months] for the gemcitabine + cisplatin arm up to the time of termination of the study).
Population: Intent-to-treat (ITT)
Measure: Count of Participants; unit: Participants
Groups:
- ORR By Central Assessment; ORR By Investigator Assessment: Infigratinib
- ORR by Central Assessment; ORR by Investigator Assessment: Gemcitabine + Cisplatin
Arm/Group | ORR By Central Assessment | ORR By Investigator Assessment | ORR by Central Assessment | ORR by Investigator Assessment
Number analyzed (Participants) | 29 | 29 | 19 | 19
Participants | 11 | 9 | 3 | 2

5. Secondary Outcome: Best Overall Response (BOR) Determined by Blinded Independent Central Assessment and the Investigator.
Description: BOR was defined as the best response a subject ever achieved after study treatment prior to crossover and any subsequent anticancer therapy, complete response (CR) and partial response (PR) were claimed only if the criteria for each were met at a subsequent time point at least 4 weeks apart. In the case of stable disease (SD), measurements must have met the SD criteria at least once post-baseline no less than 6 weeks from the randomization date.
Time Frame: as for outcome 4
Population: ITT
Measure: Count of Participants; unit: Participants
Groups:
- BOR By Central Assessment; BOR By Investigator Assessment: Infigratinib (BGJ398) 125 mg orally daily, 3 weeks on, 1 week off.
- BOR by Central Assessment; BOR by Investigator Assessment: Gemcitabine + Cisplatin Gemcitabine: Gemcitabine 1000 mg/m2 IV D1 and D8 for a 21-day cycle.
  Cisplatin: Cisplatin 25 mg/m2 IV D1 and D8 for a 21-day cycle.
Arm/Group | BOR By Central Assessment | BOR By Investigator Assessment | BOR by Central Assessment | BOR by Investigator Assessment
Number analyzed (Participants) | 29 | 29 | 19 | 19
Participants
  Confirmed complete response | 0 | 0 | 0 | 0
  Confirmed partial response | 11 | 9 | 3 | 2
  Stable disease | 14 | 19 | 11 | 12
  Progressive disease | 2 | 0 | 2 | 3
  Not done | 2 | 1 | 3 | 2

6. Secondary Outcome: Duration of Response (DOR) Determined by Blinded Independent Central Assessment and the Investigator.
Description: DOR is defined as the time from initiation of confirmed partial response (PR) or confirmed complete response (CR) to the time of confirmed progressive disease (PD) or death. If subjects do not reach PD or death before crossover, the DOR is censored at the last valid tumor assessment before crossover.
Time Frame: as for outcome 4
Population: ITT.
Measure: Median (95% Confidence Interval); unit: Months
Groups:
- DOR By Central Assessment; DOR By Investigator Assessment: Infigratinib (BGJ398) 125 mg orally daily, 3 weeks on, 1 week off.
- DOR by Central Assessment; DOR by Investigator Assessment: Gemcitabine + Cisplatin Gemcitabine: Gemcitabine 1000 mg/m2 IV D1 and D8 for a 21-day cycle.
  Cisplatin: Cisplatin 25 mg/m2 IV D1 and D8 for a 21-day cycle.
Arm/Group | DOR By Central Assessment | DOR By Investigator Assessment | DOR by Central Assessment | DOR by Investigator Assessment
Number analyzed (Participants) | 29 | 29 | 19 | 19
Months | 5.59 [3.71 to NA] — DOR is an event driven endpoint. The number of events required to assess the DOR could not be calculated due to early termination of the study. | 7.52 [3.71 to NA] — DOR is an event driven endpoint. The number of events required to assess the DOR could not be calculated due to early termination of the study. | NA [3.94 to NA] — DOR is an event driven endpoint. The number of events required to assess the DOR could not be calculated due to early termination of the study. | NA [8.08 to NA] — DOR is an event driven endpoint. The number of events required to assess the DOR could not be calculated due to early termination of the study.

7. Secondary Outcome: Disease Control Rate (DCR=PR+CR+SD) Determined by Blinded Independent Central Assessment and the Investigator.
Description: DCR is defined as the proportion of subjects with a best overall response (BOR) of either confirmed partial response (PR), confirmed complete response (CR) or stable disease (SD) or non-CR/non-PD before crossover.
Time Frame: as for outcome 4
Population: ITT
Measure: Count of Participants; unit: Participants
Groups:
- DCR By Central Assessment; DCR By Investigator Assessment: Infigratinib (BGJ398) 125 mg orally daily, 3 weeks on, 1 week off.
- DCR by Central Assessment; DCR by Investigator Assessment: Gemcitabine + Cisplatin Gemcitabine: Gemcitabine 1000 mg/m2 IV D1 and D8 for a 21-day cycle.
  Cisplatin: Cisplatin 25 mg/m2 IV D1 and D8 for a 21-day cycle.
Arm/Group | DCR By Central Assessment | DCR By Investigator Assessment | DCR by Central Assessment | DCR by Investigator Assessment
Number analyzed (Participants) | 29 | 29 | 19 | 19
Participants | 25 | 28 | 14 | 14

8. Secondary Outcome: Number of Participants With Adverse Events (AEs)
Description: Safety analyses were performed for subjects in the safety analysis population for each group. Unless otherwise specified, summaries were provided only for the on-treatment safety assessments, which are the assessments occurring or taken during the on-treatment period
Time Frame: From baseline to last dose date of study treatment + 30 days (an average of 7.5 months for the infigratinib arm and 5 months for the gemcitabine + cisplatin arm).
Population: Safety
Measure: Count of Participants; unit: Participants
Arm/Group | Infigratinib (BGJ398) 125 mg | Gemcitabine + Cisplatin
Number analyzed (Participants) | 29 | 17
Participants | 29 | 17

9. Secondary Outcome: Number of Participants With Serious Adverse Events (SAEs)
Description: as for outcome 8
Time Frame: as for outcome 8
Population: Safety
Measure: Count of Participants; unit: Participants
Arm/Group | Infigratinib (BGJ398) 125 mg | Gemcitabine + Cisplatin
Number analyzed (Participants) | 29 | 17
Participants | 10 | 0

ADVERSE EVENTS:
Time Frame: From the the time of the first administration of study treatment through 30 days after their last dose.
Description: Treatment-emergent adverse events (TEAEs) includes any AE that have onset on or after the first study treatment, and before or on either: (1) the date of data cutoff if subject was ongoing the initial study treatment; (2) the earlier of the date of last study treatment +30 days or the date of crossover if the subject received infigratinib in crossover.
Arm/Group | Infigratinib (BGJ398) 125 mg | Gemcitabine + Cisplatin
All-Cause Mortality (participants affected / at risk) | 0/29 | 0/17
Serious Adverse Events (participants affected / at risk) | 10/29 | 0/17
Other Adverse Events (participants affected / at risk) | 29/29 | 17/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Infigratinib (BGJ398) 125 mg (N=29) | Gemcitabine + Cisplatin (N=17)
Eye pain (Eye disorders) | 1 | 0
Stomatitis (Gastrointestinal disorders) | 2 | 0
Dysphagia (Gastrointestinal disorders) | 1 | 0
Fatigue (General disorders) | 1 | 0
COVID-19 (Infections and infestations) | 2 | 0
Sepsis (Infections and infestations) | 1 | 0
Calciphylaxis (Metabolism and nutrition disorders) | 1 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 0
Hyperphosphataemia (Metabolism and nutrition disorders) | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0
Hypercalcaemia of malignancy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Dizziness (Nervous system disorders) | 1 | 0
Erythema nodosum (Skin and subcutaneous tissue disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Infigratinib (BGJ398) 125 mg (N=29) | Gemcitabine + Cisplatin (N=17)
Anaemia (Blood and lymphatic system disorders) | 5 | 7
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 3
Leukocytosis (Blood and lymphatic system disorders) | 0 | 2
Neutropenia (Blood and lymphatic system disorders) | 0 | 5
Tinnitus (Ear and labyrinth disorders) | 1 | 2
Hypoacusis (Ear and labyrinth disorders) | 0 | 2
Dry eyes (Eye disorders) | 11 | 1
Keratitis (Eye disorders) | 4 | 0
Lacrimation increased (Eye disorders) | 3 | 0
Punctate keratitis (Eye disorders) | 3 | 0
Blepharitis (Eye disorders) | 2 | 1
Cataract (Eye disorders) | 2 | 0
Chorioretinopathy (Eye disorders) | 2 | 1
Eye pain (Eye disorders) | 2 | 0
Ocular hyperaemia (Eye disorders) | 2 | 0
Retinopathy (Eye disorders) | 2 | 0
Vision blurred (Eye disorders) | 1 | 1
Age-related macular degeneration (Eye disorders) | 0 | 1
Eye discharge (Eye disorders) | 0 | 1
Retinal detachment (Eye disorders) | 0 | 1
Subretinal fluid (Eye disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 14 | 4
Diarrhoea (Gastrointestinal disorders) | 13 | 5
Stomatitis (Gastrointestinal disorders) | 10 | 0
Abdominal pain (Gastrointestinal disorders) | 8 | 3
Dry mouth (Gastrointestinal disorders) | 8 | 0
Nausea (Gastrointestinal disorders) | 7 | 11
Abdominal pain upper (Gastrointestinal disorders) | 4 | 1
Vomiting (Gastrointestinal disorders) | 4 | 4
Dysphagia (Gastrointestinal disorders) | 3 | 0
Dyspepsia (Gastrointestinal disorders) | 2 | 0
Haemorrhoids (Gastrointestinal disorders) | 2 | 1
Mouth ulceration (Gastrointestinal disorders) | 2 | 0
Odynophagia (Gastrointestinal disorders) | 2 | 0
Aphthous ulcer (Gastrointestinal disorders) | 1 | 1
Ascites (Gastrointestinal disorders) | 1 | 2
Abdominal distension (Gastrointestinal disorders) | 0 | 2
Anal pruritus (Gastrointestinal disorders) | 0 | 1
Flatulence (Gastrointestinal disorders) | 0 | 1
Salivary hypersecretion (Gastrointestinal disorders) | 0 | 1
Fatigue (General disorders) | 12 | 8
Mucosal inflammation (General disorders) | 5 | 0
Asthenia (General disorders) | 4 | 5
Oedema peripheral (General disorders) | 3 | 5
Peripheral swelling (General disorders) | 0 | 2
Pyrexia (General disorders) | 2 | 5
Pain (General disorders) | 1 | 1
Hyperthermia (General disorders) | 0 | 1
Oedema (General disorders) | 0 | 1
Paronychia (Infections and infestations) | 8 | 1
COVID-19 (Infections and infestations) | 4 | 4
Urinary tract infection (Infections and infestations) | 4 | 0
Cellulitis (Infections and infestations) | 2 | 0
Sepsis (Infections and infestations) | 2 | 0
Influenza (Infections and infestations) | 0 | 1
Bronchitis (Infections and infestations) | 0 | 1
Fungal skin infection (Infections and infestations) | 0 | 1
Injection site infection (Infections and infestations) | 0 | 1
Oral candidiasis (Infections and infestations) | 0 | 1
Contusions (Injury, poisoning and procedural complications) | 2 | 0
Hand fracture (Injury, poisoning and procedural complications) | 0 | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 1
Alanine aminotransferase increased (Investigations) | 8 | 1
Aspartate aminotransferase increased (Investigations) | 6 | 0
Weight decreased (Investigations) | 6 | 2
Lipase increased (Investigations) | 5 | 0
Blood alkaline phosphatase increased (Investigations) | 3 | 1
Amylase increased (Investigations) | 2 | 0
Lymphocyte count decreased (Investigations) | 1 | 1
Platelet count decreased (Investigations) | 1 | 2
Transaminases increased (Investigations) | 1 | 1
Blood creatinine increased (Investigations) | 0 | 4
Blood lactate dehydrogenase increased (Investigations) | 0 | 1
Blood sodium decreased (Investigations) | 0 | 1
Electrocardiogram T wave inversion (Investigations) | 0 | 1
Gamma-glutamyltransferase increased (Investigations) | 0 | 1
Heart rate decreased (Investigations) | 0 | 1
Intraocular pressure increased (Investigations) | 0 | 1
Neutrophil count decreased (Investigations) | 0 | 4
White blood cell count decreased (Investigations) | 0 | 2
Hyperphosphataemia (Metabolism and nutrition disorders) | 26 | 0
Decreased appetite (Metabolism and nutrition disorders) | 12 | 5
Hypophosphataemia (Metabolism and nutrition disorders) | 12 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 7 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 7 | 2
Hyponatraemia (Metabolism and nutrition disorders) | 3 | 2
Gout (Metabolism and nutrition disorders) | 0 | 1
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 2 | 2
Hypovolaemia (Metabolism and nutrition disorders) | 2 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 2
Groin pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 11 | 4
Myalgia (Musculoskeletal and connective tissue disorders) | 6 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 6 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 5 | 5
Muscle spasms (Musculoskeletal and connective tissue disorders) | 3 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 3 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Hypercalcaemia of malignancy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Ataxia (Nervous system disorders) | 0 | 1
Neuropathy peripheral (Nervous system disorders) | 0 | 2
Polyneuropathy (Nervous system disorders) | 0 | 1
Somnolence (Nervous system disorders) | 0 | 1
Tremor (Nervous system disorders) | 0 | 1
Dysgeusia (Nervous system disorders) | 6 | 1
Headache (Nervous system disorders) | 6 | 2
Dizziness (Nervous system disorders) | 4 | 2
Paraesthesia (Nervous system disorders) | 1 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 1 | 2
Insomnia (Psychiatric disorders) | 0 | 2
Anxiety (Psychiatric disorders) | 2 | 0
Haematuria (Renal and urinary disorders) | 0 | 1
Pollakiuria (Renal and urinary disorders) | 0 | 1
Renal impairment (Renal and urinary disorders) | 0 | 1
Dysuria (Renal and urinary disorders) | 0 | 1
Amenorrhoea (Reproductive system and breast disorders) | 0 | 1
Menorrhagia (Reproductive system and breast disorders) | 0 | 1
Metrorrhagia (Reproductive system and breast disorders) | 0 | 2
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 5 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 4 | 5
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 12 | 1
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 12 | 0
Nail disorder (Skin and subcutaneous tissue disorders) | 6 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 5 | 1
Onycholysis (Skin and subcutaneous tissue disorders) | 4 | 0
Onychomadesis (Skin and subcutaneous tissue disorders) | 4 | 0
Skin fissures (Skin and subcutaneous tissue disorders) | 3 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2 | 0
Nail discolouration (Skin and subcutaneous tissue disorders) | 2 | 0
Nail dystrophy (Skin and subcutaneous tissue disorders) | 2 | 0
Onychalgia (Skin and subcutaneous tissue disorders) | 2 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 2
Rash (Skin and subcutaneous tissue disorders) | 2 | 1
Skin disorder (Skin and subcutaneous tissue disorders) | 2 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 1
Flushing (Vascular disorders) | 0 | 1
Phlebitis (Vascular disorders) | 0 | 2
Hypotension (Vascular disorders) | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-07-27): https://cdn.clinicaltrials.gov/large-docs/02/NCT03773302/Prot_000.pdf
  • Statistical Analysis Plan (2023-03-08): https://cdn.clinicaltrials.gov/large-docs/02/NCT03773302/SAP_001.pdf